CLINICAL TRIAL: NCT03117322
Title: Efficacy of the Supplementation With a Symbiotic, a Prebiotic and a Probiotic to Produce a Beneficial Effect on the Intestinal Microbiota and on the Characteristics of Feces in Children With Cerebral Palsy (CP) and Chronic Constipation
Brief Title: Synbiotic, Prebiotics and Probiotics in Children With Cerebral Palsy and Constipation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Andrea Garcia Contreras (Other)
Responsible Party: Sponsor-Investigator, Andrea Garcia Contreras, Principal investigator, Hospital Civil Juan I. Menchaca
Organization: Hospital Civil Juan I. Menchaca (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 0167/17
Record Dates: First submitted 2017-04-10; First posted 2017-04-17 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-04

CONDITIONS: Cerebral Palsy; Chronic Constipation
Keywords: cerebral palsy; children; chronic constipation; synbiotic; prebiotics; probiotics; agave inulin; microbiota
MeSH Terms: conditions — Cerebral Palsy | interventions — maltodextrin; Sunflower Oil

STUDY DESIGN:
Intervention Model Description: Three interventions in parallel against a control group
Who Masked: Participant, Care Provider, Investigator
Masking Description: pediatric neurologist and laboratory staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Synbiotic (Experimental): Each participant will receive the next:
  1. agave inulin (4 g) in powder
  2. Lactobacillus reuteri DSM 17938 (1 x 10^8 cfu) in 5 drops daily, once a day for four weeks.
  Interventions: Biological: agave inulin; Biological: Lactobacillus reuteri DSM 17938
- Probiotic (Experimental): Lactobacillus reuteri DSM 17938 (1 x 10^8 cfu) in 5 drops and maltodextrin (4 g) in powder daily, once a day for four weeks.
  Interventions: Biological: Lactobacillus reuteri DSM 17938; Other: maltodextrin
- Prebiotic (Experimental): agave inulin (4 g) in powder and an oil mix (sunflower oil and medium chain triglyceride oil) in 5 drops daily, once a day for four weeks.
  Interventions: Biological: agave inulin; Other: Oil mix (medium chain triglycerides and sunflower oil)
- Placebo (Placebo Comparator): maltodextrin (4 g) in powder and an oil mix (sunflower oil and medium chain triglyceride oil) in 5 drops daily, once a day for four weeks.
  Interventions: Other: maltodextrin; Other: Oil mix (medium chain triglycerides and sunflower oil)

INTERVENTIONS:
Biological: agave inulin — Duration: four weeks Dosage: powder 4 g/d
  Arms: Prebiotic; Synbiotic
Biological: Lactobacillus reuteri DSM 17938 — Duration: four weeks Dosage: 5 drops/d
  Arms: Probiotic; Synbiotic
Other: maltodextrin — Duration: four weeks Dosage: powder 4 g/d
  Arms: Placebo; Probiotic
Other: Oil mix (medium chain triglycerides and sunflower oil) — Duration: four weeks Dosage: 5 drops/d
  Arms: Placebo; Prebiotic

SUMMARY:
Randomized double blind controlled clinical trial. Participants will be enrolled at the New Civil Hospital of Guadalajara "Dr. Juan I. Menchaca" during the period from May 2017 to July 2018, from six to 59 months of either sex. The duration of each participant in the study will be of four weeks. Each participant will be randomized assigned to any of the different study groups: synbiotic, prebiotic, probiotic or placebo. Hypothesis: The efficacy of supplementation with a symbiotic, a prebiotic and a probiotic differs in its beneficial effect on the intestinal microbiota and the characteristics of feces in children with CP and chronic constipation.

DETAILED DESCRIPTION:
All the data registered in the case report forms will be monitored by the responsible party. This person will be monitoring each procedure during the study.

All the data in the case report forms will be obtained from the information obtained from the legal caregiver or the parents of the child and/or from the medical and electronic records and calls to the parents or legal caregivers and will be introduced daily in the Statistical Package for the Social Scienses (SPSS) program version 21. The responsible party will have access to this database and will verify the information.

Plan for missing data. In case that we have some missing variables, we will call the parents or legal caregiver of the children if it is about the data of the child. In case of missing data, unavailable or non-reported variable and it is not possible to compare the initial vs final phases, the subject will be excluded from the study. In case of finding an out-of-range laboratory results we will repeat the test. If we have some missing data from the subject but we can analyze other results from the same subject, it will not be excluded.

Standard Operating Procedures to address registry operations and analysis activities, such as patient recruitment, data collection, data management, data analysis, reporting for adverse events, and change management. Patients will be recruited from the nutrition and neurology outpatient at the New Hospital Civil of Guadalajara. We will apply a standardized questionnaire to the parents or legal caregivers to assure that the subject could be eligible to the study. Once all the inclusion criteria are fulfilled then another questionnaire or case report form will be filled. The informed consent will be explained and given to the parents or legal caregivers of the child for sign. An external person will be chose to assign randomly (by envelops) the subjects to each group. This person will provide the study product and the diaries to the parents or legal caregivers. Data from the case reports forms will be captured by the principal investigator and monitored by the responsible party. Te adverse events will be reported by phone calls during the four weeks (two to three phone calls in a week). To analyze the information, the SPSS program version 21 will be used.

Sample size. The sample size was calculated according to the next formula:

n= K (σ12 + σ22)/ (μ1 - μ2) 2 = 6.2 (1.12 + 0.62)/ (4.01 - 2.8) n= 7 + 3 (30% probability of exclusion) = 10 children for each group, total subjects in the study: 40.

α= 0.05 β= 0.20 Data was obtained from the study of Indrio F, et al (2014) 18 with the number of evacuation.

Sampling system. Simple random sample by means of closed envelopes with a figure inside. We will have 40 envelopes closed, 10 of them will have a circle, 10 a triangle, 10 a star and 10 a heart. They will be put into a box; this will be rotated five times before taking an envelope. Randomly, a person outside the study will take an envelope, will see the chosen figure and will write it down in the register.

Statistical analysis. First stage. Shapiro Wilk test will be performed to see the distribution of the data. Descriptive statistics: mean, standard deviation, percentages and frequencies will be performed. Second stage. Analytical statistics: Intra-groups: Student's T test for dependent samples for parametric data or the Wilcoxon test for non-parametric data. Chi square for analysis of qualitative data. Inter-groups: One-way ANOVA with post hoc (Bonferroni) tests. If the data are not parametric, Kruskal-Wallis and if it is significant, Mann Whitney's U will be performed as post hoc. Third stage. Linear regression and logistic regression will be performed.

Ethical considerations. Parents or legal representatives of the child will be informed about the study, requesting their signature for consent. Human research guidelines will be respected according to "good clinical practice". The protocol will be submitted to the Bioethics Committee of the New Civil Hospital of Guadalajara and the University of Guadalajara. Care will be taken to respect the recommendations of the Helsinki Declaration in its last correction made during the 64th Annual Assembly organized by the World Medical Association (2013).

ELIGIBILITY:
Inclusion Criteria:

* Participants attending the outpatient of nutrition and/or pediatric neurology with cerebral palsy diagnosed and confirmed by a pediatric neurologist, and that belong to levels IV or V of the Gross Motor Function Classification System (GMFCS).
* Participants with constipation according to the Rome IV criteria.
* Signed informed consent by one of the child's parents or legal guardians

Exclusion Criteria:

* Refusal to continue in the study
* Use of antibiotics during the study, consumption of laxatives, food fibers, lactulose, magnesia or products containing probiotics, prebiotics or both as infant formulas (NOTE: Glycerin suppositories will only be allowed when there is no evacuation for more than five days).
* Omission of administration of the required dose of symbiotic, prebiotic, probiotic or placebo and/or administered with an unspecified frequency (compliance <95%)
* Adverse effects not related to the agent of study.

Ages: 6 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Change in the composition of the microbiota (firmicutes, bifidobacteria and lactobacilli) | change from baseline bacteria composition at four weeks
  species/g
change in consistency of feces | change from baseline consistency at four weeks
  Bristol scale
change in potential of hydrogen (pH) of feces | Change from baseline pH at four weeks
  pH scale
change in frequency of evacuations | change from baseline frequency at four weeks
  evacuations per week

SECONDARY OUTCOMES:
change in the concentration of short chain fatty acids in feces | Change from baseline concentration at four weeks
  millimoles (mM)

OTHER OUTCOMES:
Change in Body weight | Change from baseline weight at four weeks
  Kg
length | Baseline
  cm
Change of Dietary fiber intake | Change from baseline dietary fiber intake at four weeks
  grams
Change of dietary Liquids | Change from baseline liquids at four weeks
  milliliters (mL)

CONTACTS AND LOCATIONS:
Overall Officials: Edgar M Vásquez-Garibay, Doctor, Principal Investigator — full time staff member at the Division of Pediatrics of the New Civil Hospital of Guadalajara
Locations (1):
- Nuevo Hospital Civil de Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ojetti V, Ianiro G, Tortora A, D'Angelo G, Di Rienzo TA, Bibbo S, Migneco A, Gasbarrini A. The effect of Lactobacillus reuteri supplementation in adults with chronic functional constipation: a randomized, double-blind, placebo-controlled trial. J Gastrointestin Liver Dis. 2014 Dec;23(4):387-91. doi: 10.15403/jgld.2014.1121.234.elr. PMID 25531996
- [Background] Indrio F, Di Mauro A, Riezzo G, Civardi E, Intini C, Corvaglia L, Ballardini E, Bisceglia M, Cinquetti M, Brazzoduro E, Del Vecchio A, Tafuri S, Francavilla R. Prophylactic use of a probiotic in the prevention of colic, regurgitation, and functional constipation: a randomized clinical trial. JAMA Pediatr. 2014 Mar;168(3):228-33. doi: 10.1001/jamapediatrics.2013.4367. PMID 24424513
- [Background] Coccorullo P, Strisciuglio C, Martinelli M, Miele E, Greco L, Staiano A. Lactobacillus reuteri (DSM 17938) in infants with functional chronic constipation: a double-blind, randomized, placebo-controlled study. J Pediatr. 2010 Oct;157(4):598-602. doi: 10.1016/j.jpeds.2010.04.066. Epub 2010 Jun 12. PMID 20542295
- [Background] Choi CH, Chang SK. Alteration of gut microbiota and efficacy of probiotics in functional constipation. J Neurogastroenterol Motil. 2015 Jan 31;21(1):4-7. doi: 10.5056/jnm14142. No abstract available. PMID 25611063
- [Background] Attaluri A, Jackson M, Valestin J, Rao SS. Methanogenic flora is associated with altered colonic transit but not stool characteristics in constipation without IBS. Am J Gastroenterol. 2010 Jun;105(6):1407-11. doi: 10.1038/ajg.2009.655. Epub 2009 Dec 1. PMID 19953090
- [Background] Elawad MA, Sullivan PB. Management of constipation in children with disabilities. Dev Med Child Neurol. 2001 Dec;43(12):829-32. doi: 10.1017/s0012162201001505. No abstract available. PMID 11769270
- [Background] Tse PW, Leung SS, Chan T, Sien A, Chan AK. Dietary fibre intake and constipation in children with severe developmental disabilities. J Paediatr Child Health. 2000 Jun;36(3):236-9. doi: 10.1046/j.1440-1754.2000.00498.x. PMID 10849223
- [Background] Del Giudice E, Staiano A, Capano G, Romano A, Florimonte L, Miele E, Ciarla C, Campanozzi A, Crisanti AF. Gastrointestinal manifestations in children with cerebral palsy. Brain Dev. 1999 Jul;21(5):307-11. doi: 10.1016/s0387-7604(99)00025-x. PMID 10413017
- [Background] Park ES, Park CI, Cho SR, Na SI, Cho YS. Colonic transit time and constipation in children with spastic cerebral palsy. Arch Phys Med Rehabil. 2004 Mar;85(3):453-6. doi: 10.1016/s0003-9993(03)00479-9. PMID 15031832
- [Background] Sullivan PB, Lambert B, Rose M, Ford-Adams M, Johnson A, Griffiths P. Prevalence and severity of feeding and nutritional problems in children with neurological impairment: Oxford Feeding Study. Dev Med Child Neurol. 2000 Oct;42(10):674-80. doi: 10.1017/s0012162200001249. PMID 11085295
- [Background] Morad M, Nelson NP, Merrick J, Davidson PW, Carmeli E. Prevalence and risk factors of constipation in adults with intellectual disability in residential care centers in Israel. Res Dev Disabil. 2007 Nov-Dec;28(6):580-6. doi: 10.1016/j.ridd.2006.08.002. Epub 2007 Mar 2. PMID 17336497
- [Background] Bohmer CJ, Taminiau JA, Klinkenberg-Knol EC, Meuwissen SG. The prevalence of constipation in institutionalized people with intellectual disability. J Intellect Disabil Res. 2001 Jun;45(Pt 3):212-8. doi: 10.1046/j.1365-2788.2001.00300.x. PMID 11422645
- [Background] Rosenbaum P. The natural history of gross motor development in children with cerebral palsy aged 1 to 15 years. Dev Med Child Neurol. 2007 Oct;49(10):724. doi: 10.1111/j.1469-8749.2007.00724.x. No abstract available. PMID 17880638